CLINICAL TRIAL: NCT01442974
Title: Assessment Of Stromal Response To Nab-Paclitaxel In Combination With Gemcitabine In Pancreatic Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Grupo Hospital de Madrid (Other)
Responsible Party: Principal Investigator, Sofia Perea, Director Clinical Trials Unit., Director Clinical Research Unit, Grupo Hospital de Madrid
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABX271-PA09EU
Record Dates: First submitted 2011-06-13; First posted 2011-09-29 (Estimated); Last update posted 2013-03-13 (Estimated); Status verified 2013-03

CONDITIONS: Pancreatic Cancer
Keywords: nab-paclitaxel; neoadjuvant treatment; SPARC; Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gemcitabine plus nab-paclitaxel (Experimental): This is a single arm study.
  Interventions: Drug: Gemcitabine plus nab-paclitaxel

INTERVENTIONS:
Drug: Gemcitabine plus nab-paclitaxel — Gemcitabine 1000mg/mq on d1,8,15 over 28 days of cycle nab-paclitaxel 125mg/mq on d1,8,15 over 28 days cycle Treatment will be administered for two cycles
  Other Names: Gemzar; 2'-deoxy-2',2''-difluorocytidine-5'-O-monophosphate; Abraxane; ABI007

SUMMARY:
Targeting tumor stroma is emerging as a strategic approach for pancreatic cancer treatment. Actually, one of the most interesting characteristics of pancreatic cancer is the dense fibrotic stroma surrounding tumor cells. Moreover, pancreatic cancer stroma seems to express a specific protein profile different from tumor cells. For example, secreted protein rich in cysteine (SPARC) is overexpressed in pancreatic tumor stroma fibroblast and downregulated in tumor cells. This characteristic is associated with poor clinical outcome.

Nab-paclitaxel, an albumin bound nano formulation of paclitaxel that targets SPARC, decreases tumor stroma density. Such effect improves drug delivery, and enhances both, nab-paclitaxel and gemcitabine, antitumor activity in nude mouse models.

Based on this pre-clinical data the investigators designed a clinical trial of nab-paclitaxel in combination with gemcitabine as neo-adjuvant treatment for pancreatic cancer patients. Fifteen, SPARC positive patients, will be enrolled in the study and treated with abraxane in combination with gemcitabine.

This is a pilot study which primary end point is evaluating the effect of Abraxane in combination with gemcitabine on tumor stroma, and the secondary end-point is correlating these changing with treatment activity.

DETAILED DESCRIPTION:
Study Phase: Pilot study to assess nab-paclitaxel in combination with gemcitabine effects on pancreatic cancer stroma and tumor metabolism.

Study Objective(s):

A) Primary end-points:

1. Evaluate the effect of nab-paclitaxel in combination with gemcitabine on tumor stroma density.
2. Evaluate the effect of nab-paclitaxel on tumor vessels formation.
3. Evaluate the effect of nab-paclitaxel on tumor metabolism.

B) Secondary end-point:

1. Evaluate combination activity in relation with changes in tumor stroma and tumor metabolic activity.

The following studies will be performed prior and after treatment administration:

* 18FDG-PET/CT scan;
* Ultrasound Elastography;
* IHC:

  1. SPARC;
  2. Microvessel Density (CD-31, VEGF-A);
  3. Stroma density (SMA and Collagen I).

Study population and Number of subject: A total of 15 pancreatic cancer patients with resectable/resectable borderline disease are expected to be enrolled.

Study design and schedule: This is a pilot study to evaluate the effect of nab-paclitaxel on tumor stroma in pancreatic cancer patients. The study will be conducted in two parts:

Part A: Patients diagnosed with resectable/resectable pancreatic cancer will be screened for SPARC expression. Fifteen, SPARC positive patients, will be enrolled in the study and treated with nab-paclitaxel in combination with gemcitabine. Patients will be treated as follow:

* nab-paclitaxel will be administered at 125 mg/m2 as intravenous (i.v.) infusion over 30 minutes;
* followed by gemcitabine 1000 mg/m2 i.v. infusion over 30 minutes;

Treatment will be delivered weekly, for 3 weeks (on day 1, 8, and 15 over 28 days cycle) followed by a week of rest, for two cycles of treatment.

Part B: At the end of treatment tumors will be surgically resected according to standard surgical procedure for the treatment of pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are 18 years or older;
* Patients with resectable/resectable borderline pancreatic cancer;
* Adequate hematopoietic, hepatic and renal function:

  * Neutrophil count > o = 1.5 x 109/L;
  * Platelet count > o = 100 x 109/L;
  * Bilirubin ≤ 1.5 x ULN;
  * AST and/or ALT ≤ 2.5 x ULN;
  * Serum creatinine ≤ 1.5 x ULN.
* Investigators must ensure that patients enrolled in the study will be available for all study procedures, including tumor biopsy, surgical treatment, and follow up.
* Investigators must ensure that patients have the ability to understand the requirements of the study and provide signed informed consent.
* Signed Informed Consent.

Exclusion Criteria:

* Active or uncontrolled infections or serious illnesses or medical conditions that could interfere with patient eligibility for treatment;
* History of any psychiatric condition that might impair patient's ability to understand or to comply with the requirements of the study or to provide informed consent;
* Concurrent anticancer therapy;
* Pregnant or breast-feeding women (documented methods of birth control are required in those with reproductive potential);
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to study drugs;
* History of life threatening reaction to gemcitabine or abraxane;
* Previous exposure to other agents or treatment procedure as radiotherapy for the treatment of pancreatic cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-01; Primary Completion 2012-01 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Effect of nab-paclitaxel on pancreatic cancer stroma, new vessel formation and tumor cell metabolism. | up to 18 months
  Primary End-point:
  1. Evaluate the effect of nab-paclitaxel in combination with gemcitabine on tumor stroma density.
  2. Evaluate the effect of nab-paclitaxel on tumor vessels formation.
  3. Evaluate the effect of nab-paclitaxel on tumor metabolism by PET-CT scan measuring pre-treatment versus post-treatment glucose uptake.

SECONDARY OUTCOMES:
Activity of nab-paclitaxel in combination with gemcitabine against PDA in relation with changes in tumor stroma and tumor metabolic activity. | up to 18 months
  To assess secondary end-point the following studies will be performed
  * 18FDG-PET/CT scan;
  * Ultrasound Elastography;
  * IHC:
    1. SPARC;
    2. Microvessel Density (CD-31, VEGF-A);
    3. Stroma density (SMA and Collagen I).

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Hidalgo, MD, PhD, Principal Investigator — Centro Integral Oncologico Clara Campal (CIOCC), Centro National Investigacion Oncologica (CNIO)
Locations (1):
- Centro Integral Oncologico Clara Campal, Madrid, Spain